CLINICAL TRIAL: NCT01139112
Title: Klebsiella Pneumoniae Necrotizing Fasciitis: Clinical and Microbiological Features
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201005034R
Record Dates: First submitted 2010-06-07; First posted 2010-06-08 (Estimated); Last update posted 2012-11-15 (Estimated); Status verified 2012-05

CONDITIONS: Necrotizing Fasciitis
Keywords: Necrotizing Fasciitis, Klebsiella Pneumoniae
MeSH Terms: conditions — Fasciitis, Necrotizing

STUDY DESIGN:
Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — K. pneumoniae strains stored at -80oC
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a retrospective descriptive study on the clinical and microbiological features of Klebsiella Pneumoniae Necrotizing Fasciitis.

DETAILED DESCRIPTION:
Background. Necrotizing fasciitis is a rapidly progressive, life-threatening infectious disease that primarily involves soft tissue. Traditionally, group A streptococcus is the major cause of this disease. In recent years, however, there are increasing case reports of necrotizing fasciitis solely caused by Klebsiella pneumoniae. There are limited data regarding clinical and microbiological features of K. pneumoniae strains causing this disease.

Methods. We plan to review the medical records of necrotizing fasciitis cases treated during 1997-2010 at National Taiwan University Hospital, and compare the clinical features of cases caused by K. pneumonia and cases caused by group A streptococcus. We also plan to retrospectively identify necrotizing fasciitis-associated K. pneumoniae strains stored at -80oC at National Taiwan University Hospital, and perform virulence-associated hypermucoviscosity phenotyping, wzy (magA locus) and rmpA genotyping, and detection of 20-kb kfu/PTS genomic region and other iron-uptake systems.

Expected Results. This study is expected to yield the following important information: (1) The prevalence of monomicrobial K. pneumoniae necrotizing fasciitis cases among all necrotizing fasciitis cases at our hospital during the study period; (2) The distinct clinical features of K. pneumoniae necrotizing fasciitis, using group A streptococcal necrotizing fasciitis as the comparison group; (3) The microbiologic characteristics of K. pneumoniae strains causing monomicrobial necrotizing fasciitis, including hypermucoviscosity phenotype, wzy (magA locus) and rmpA genotype, and the presence of iron-uptake systems.

ELIGIBILITY:
Inclusion Criteria:

* Definitive diagnosis of necrotizing fasciitis depends on intra-operative findings characterized by a lack of resistance to blunt dissection of the normally adherent fascia, presence of necrotic fascia, and purulent malodorous discharge. Pathological findings of the involved fascia typically show neutrophils and bacterial clumps infiltrating between collagen bundles of with focal necrosis.

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Necrotizing fasciitis cases treated during 1997-2010 at National Taiwan University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 134 (Actual)
Dates: Start 2009-07; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chi-Tai Fang, MD, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taipei, Taiwan